CLINICAL TRIAL: NCT00697034
Title: Effects of Capsaicin on the Structure, Distribution, and Function of Cutaneous Small Nerve Fibers in Psoriatic Skin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of qualified and willing volunteers.
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-467
Record Dates: First submitted 2008-06-09; First posted 2008-06-13 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Capsaicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- 1 (Experimental): Study subjects will be patients with chronic plaque-type psoriasis
  Interventions: Drug: Capsaicin

INTERVENTIONS:
Drug: Capsaicin — natural alkaloid derived from hot chili peppers and activates vanilloid receptors that are also activated by endogenous cannabinoid anandamide applied three times daily

SUMMARY:
The purpose of this research study is to examine the role of nerves in the skin in psoriasis and to better understand the effects of capsaicin in psoriasis.In this study, capsaicin will be compared to a moisturizer (aquaphor ointment).

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women who are 18 years of age or older.
* Diagnosis of plaque-type psoriasis is required to be confirmed by clinical criteria.
* Subjects must be in general good health with no other skin disease, disease state or physical condition which would impair evaluation of psoriasis or which would increase their health risk by study participation.
* Subjects must be willing to receive topical capsaicin weekly for 6 weeks and must be willing to undergo 3mm punch biopsies at baseline and at week 6.
* Subjects may not receive any systemic therapies during the study.
* Subjects are required to complete a 4 week washout period from any systemic medication and/or phototherapy prior to enrolling in the study.
* Stable use of moisturizers will be allowed provided that use has been stable for at least 14 days.
* Women of child bearing age will be required to have a negative pregnancy test in order to enroll in the study and will be required to maintain adequate birth control throughout the study.

Exclusion Criteria:

* Subjects who are unable to complete the required measures.
* Subjects diagnosed with other skin diseases that would affect the measurement of cutaneous blood flow.
* Subjects with any history of any disease associated with neuropathy, including diabetes, alcoholism, uremia, HIV infection, hypothyroidism, or cancer chemotherapy.
* Subjects who are currently enrolled in any investigational study in which the subject is receiving any type of drug, biologic, or non-drug therapy and subjects undergoing treatment with another investigational drug or approved therapy for investigational use within 28 days prior to investigational drug administration.
* Subjects who have used any topical therapy for psoriasis or other skin diseases in the past 7 days.
* Subjects receiving any of the following treatments or agents within the 28 days prior to investigational drug administration will be excluded: systemic retinoids, systemic steroids, methotrexate, cyclosporine, azathioprine, thioguanine, etanercept, efalizumab, infliximab, adalimumab or mofetil or other systemic immunosuppressant, and phototherapy, including Ultraviolet B (UVB) and Psoralen + Ultraviolet A (PUVA).
* Subjects with a known allergy to capsaicin.
* Children less than 18 years of age.
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-06; Primary Completion 2007-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To assess the effect of capsaicin on small nerve fiber function in psoriasis | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Gil Yosipovitch, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States